CLINICAL TRIAL: NCT07027137
Title: The Influence of Local Antibiotic Therapy on the Outcomes Following Periodontal Regeneration Procedures.
Acronym: ANBperio
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniBial2; R-I-002/403/2019 (Other: University of Bialystok)
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Periodontitis; Periodontal Diseases
Keywords: periodontitis; periodontal regeneration; local antibiotics
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: The study group consisted of 20 people participants who underwent the SRP procedure (scaling and root planing) performed with the subsequent application of local antibiotics (10% doxycycline) into periodontal pockets at the site of the planned surgical intervention, while in the control group SRP was performed alone. Two weeks after SRP, the M-MIST/MIST procedure was performed in both the test and control groups with the use of enamel matrix derivative (EMD). All surgical interventions were performed under local anesthesia (Septanest, Septodont, Paris, France). After intrabony defect exposure the granulation tissue was excised using the hand instruments (Gracey currettes (SMS), Hu-Friedy, Chicago, IL, USA), the root surface was conditioned with 24% EDTA (PrefGel®, Straumann, Switzerland) and defect was filled with enamel matrix derivative (Emdogain®, Straumann, Switzerland). Once procedure was completed, the mucoperiosteal flap was repositioned and stabilized with sutures.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRP+SURG (Experimental): In the control group (20 subjects) SRP was performed alone. After two weeks regeneration procedure was performed.
  Interventions: Procedure: SRP+SURG
- SRP+ANB+SURG (Experimental): The test group consisted of 20 people participants who underwent the SRP procedure with local antibiotic application into the pocket was performed. After two weeks regeneration procedure was performed.
  Interventions: Drug: SRP+ANB+SURG

INTERVENTIONS:
Drug: SRP+ANB+SURG — SRP (scaling and root planing) with ANB (local antibiotic application- 10%doxycycline) and SURG (regeneration procedure according to MIST/M-MIST)
  Arms: SRP+ANB+SURG
Procedure: SRP+SURG — SRP (scaling and root planing) and SURG (regeneration procedure according to MIST/M-MIST)
  Arms: SRP+SURG

SUMMARY:
Assessmnet of the influence of local antibiotic therapy on the clinical, radiological, microbiological parameters and the inflammation mediators levels in the gingival crevicular fluid (GCF) following periodontal regeneration procedures in patients with periodontitis.

DETAILED DESCRIPTION:
Forty generally healthy adults diagnosed with stage III periodontitis were randomly divided into two groups. In the test group, SRP was performed with the subsequent application of local antibiotics (10% doxycycline) into periodontal pockets at the site of the planned surgical intervention, while in the control group SRP was performed alone. Two weeks after, on the day of the surgical treatment, the M-MIST/MIST procedure was performed in both the test and control groups with the use of enamel matrix derivative (EMD). Clinical examination was performed before and 6 and 12 months after treatment. For radiological measurements RVG was performed. For inflammation mediators levels determination in GCF samples ELISA method will be used. For microbiological assessments Real Time PCR method will be used.

ELIGIBILITY:
Inclusion Criteria:

-presence of an intrabony defect, with a pocket depth (PD) ≥ 6 mm and a radiological defect depth of ≥3 mm and width of ≥2 mm;

Exclusion Criteria:

* periodontal treatment within 3 months prior to the study;
* antibiotic therapy within 3 months prior to the study;
* smoking; presence of systemic diseases affecting periodontal healing, i.e.: immunosuppressive diseases, diabetes, osteoporosis, AIDS, hypertension treated with calcium channel blockers;
* use of steroids or other immunosuppressive drugs;
* pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the influence of local antibiotic therapy on the clinical, outcomes following periodontal regeneration procedures. | up to 12 months after treatment procedure
  PD (Pocket Depth) reduction- measured from the gingival margin to the bottom of the sulcus (mm) CAL (Clinical Attachment Level) gain- measured from the cemento-enamel junction to the bottom of the sulcus (mm)

SECONDARY OUTCOMES:
Assessment of the influence of local antibiotic therapy on the radiological outcomes following periodontal regeneration procedures. | up to 12 months after treatment procedure
  RIDW- (radiological intrabony defect width)- measured from bone crest to the root surface (mm) RIDD - (radiologial intrabony defect depth) - measured from bone crest to the bottom of the defect (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Integrated Dentistry, Medical University of Białystok, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
IPD cannot be transferred to other people due to GDPR